CLINICAL TRIAL: NCT05534711
Title: Family Stress Study: A Longitudinal Observational Study Examining Chronic Stress and Weight Gain Pathways in Young Children.
Brief Title: The Family Stress Study - Chronic Stress and Child Adiposity: Testing a Bio-behavioural Model
Status: Active, not recruiting | Type: Observational
Sponsor: University of Guelph (Other)
Collaborators: McMaster University (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Jess Haines, Dr. Jess Haines, University of Guelph
Other Study IDs: FSS
Record Dates: First submitted 2022-07-15; First posted 2022-09-09 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Pediatric Obesity; Mental Health Wellness 1
Keywords: Chronic stress; Child obesity; Household chaos; Parental depression; COVID19; Child mental health
MeSH Terms: conditions — Pediatric Obesity; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The Family Stress Study is following families with young children in Guelph, Hamilton and surrounding areas over 3 years to understand how chronic stress impacts children's weight gain over time and how this association is mediated by alterations in children's cortisol production and weight-related behaviours.

DETAILED DESCRIPTION:
The Family Stress Study is a longitudinal observational study designed to examine behavioural and biological pathways through which exposure to chronic stress may impact excess weight gain in young children.

This study will examine whether exposure to chronic stressors, i.e., household chaos, negative life events, food insecurity, and parental depression, is directly associated with higher weight gain among children. This study will also examine whether alterations in children's cortisol production and weight-related behaviours, i.e., dietary intake, eating behaviour, physical activity, sedentary behaviours and sleep, mediate the stress-weight gain link in young children. This research will also identify whether the quality of caregiver relationships, child sex, family social support, family social connection, or caregiver education moderate the pathways linking stress and excess weight gain.

To achieve our aims, 360 children aged 2 to 6 years from families in the Guelph and Hamilton areas will be recruited to examine key behavioural and biological pathways through which exposure to chronic stress may impact weight gain. Our study will also examine the impact of chronic stress on children's mental health, which is a secondary outcome of our study. Understanding which sources of stress and the key behaviours that have the greatest impact on obesity risk among chronically stressed children will aid in the development of effective obesity prevention interventions for specific families.

Additionally, this study is well-poised to examine how family stressors during the COVID-19 pandemic influenced children's health behaviours and resulting weight outcomes. Further examination of COVID-19-related stressors, i.e., quarantine or illness due to COVID-19, employment in essential services, general stress, food insecurity, financial insecurity and employment change due to COVID-19, impact cortisol levels and health behaviours and resulting weight outcomes in children. We will also examine how factors such as family social connection or social support, may moderate the impact of the stressors due to COVID-19 on child health. This information will guide strategies to support families in the post-COVID-19 context.

ELIGIBILITY:
Inclusion Criteria:

* Families are eligible to participate if they have at least 1 adult caregiver responsible for the care of a child aged 2-6 years at the time of enrollment (target age group for the study);
* Families must live in the Guelph (i.e.: Wellington County- includes Guelph, Rockwood, Fergus, Elora, Mount Forest, Puslinch, Cambridge, Kitchener, Waterloo) or Hamilton (i.e.: Municipality of Hamilton-Wentworth - includes Hamilton, Ancaster, Dundas, Flamborough, Glanbrook, Stoney Creek as well as Burlington) areas and must not be planning to move outside of these areas within three years;

Exclusion Criteria:

* Language - The participating caregiver must be fluent in English since all study communications and survey questions are in English;
* Participation in the Guelph Family Health Study (GFHS) - families previously or currently participating in the GFHS will be excluded as the GFHS provided intervention that may bias the results of the current study;
* Child custody - The participating caregiver must have at least 50% shared custody of their child (to allow for separated/divorced families to participate ensuring caregivers' reports of family-level stressors are relevant for the child);
* Health conditions of the children impacting cortisol production, obesity and/or growth/body composition - Hair sample cortisol, fat mass and growth measurements would be affected by these conditions (e.g. Cushing's Disease, Prader Willi Syndrome, untreated thyroid disease);
* Children taking steroid medications including oral or inhaled corticosteroids - Hair sample cortisol measurements would be affected by the use of steroid medications;
* Children taking medications for ADHD (attention deficit hyperactivity disorder), antidepressants or antipsychotic medications - These medications can affect body composition;
* Children born before 34 weeks gestation - Body composition and growth can be affected for children born before 34 weeks.

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Family: For this study, we define family as caregivers and their oldest eligible child who is 2-6 years old. Families can have one or many caregivers. Up to two caregivers from each family can register to take part in this study;
  Caregiver(s): We define caregivers as the main adults who regularly provide direct care for children of a family. Examples of caregivers include parents (can be biological, related, adoptive or foster if living with the child full time), grandparents, aunts and uncles. One participating caregiver must have at least 50% custody or 50% legal guardianship of the oldest eligible child who is 2-6 years old.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-07-09 (Actual); Primary Completion 2027-05-30 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
Child Body Composition - Waist Circumference | Year 2 (T3)
  Child waist circumference in cm
Child Body Composition - Child BMIz Score | Year 2 (T3)
  Child BMIz score in kg/m2 - combined weight height, age, sex

SECONDARY OUTCOMES:
Mental health in children | Year 5 (T4)
  Mental health outcomes in children using survey measures of stress, adverse life events, and psychosocial problems.

CONTACTS AND LOCATIONS:
Overall Officials: Jess Haines, PhD, Principal Investigator — University of Guelph
Locations (2):
- Canada (2):
  - University of Guelph, Guelph, Ontario
  - McMaster University, Hamilton, Ontario

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Pare SM, Gunn E, Morrison KM, Miller AL, Duncan AM, Buchholz AC, Ma DWL, Tremblay PF, Vallis LA, Mercer NJ, Haines J. Testing a Biobehavioral Model of Chronic Stress and Weight Gain in Young Children (Family Stress Study): Protocol and Baseline Demographics for a Prospective Observational Study. JMIR Res Protoc. 2024 Jun 20;13:e48549. doi: 10.2196/48549. PMID 38900565